CLINICAL TRIAL: NCT06596395
Title: Effect of Acute Caffeine and Beetroot Juice Intake on Strength, Power, and Muscular Endurance Based on Circadian Rhythms.
Brief Title: Effect of Acute Caffeine and Beetroot Juice Intake on Strength, Power, and Muscular Endurance
Acronym: CAF+BJ
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alcala (Other)
Responsible Party: Principal Investigator, Alberto Pérez-López, Principal Investigator, University of Alcala
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Other
Other Study IDs: CEIP/2023/4/093
Record Dates: First submitted 2024-09-06; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Dietary Supplements; Caffeine; Nitrates; Sports Performance; Resistance Exercise

STUDY DESIGN:
Intervention Model Description: Triple-blind, cross-over, randomized controlled-trial
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Caffeine + Beetroot Juice (Experimental): 70 mL of concentrated NO3--rich (BJ, 6.5 mmol NO3-) + 3 mg/kg of caffeine
  Interventions: Dietary Supplement: Acute caffeine and beetroot juice
- Beetroot Juice (Experimental): 70 mL of concentrated NO3--rich (BJ, 6.5 mmol NO3-) + 3 mg/kg of placebo (maltodextrin)
  Interventions: Dietary Supplement: Acute beetroot juice
- Caffeine (Experimental): 70 mL of NO3--depleted (BJ, 0.04 mmol NO3-) + 3 mg/kg of caffeine
  Interventions: Dietary Supplement: Acute caffeine
- Placebo (Placebo Comparator): 70 mL of NO3--depleted (BJ, 0.04 mmol NO3-) + 3 mg/kg of placebo (maltodextrin)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Acute caffeine and beetroot juice — Combined effect of beetroot juice and caffeine intake on muscular strength, power and endurance performance
  Arms: Caffeine + Beetroot Juice
Dietary Supplement: Acute caffeine — single effect of caffeine intake on muscular strength, power and endurance performance
  Arms: Caffeine
Dietary Supplement: Acute beetroot juice — single effect of beetroot juice intake on muscular strength, power and endurance performance
  Arms: Beetroot Juice
Dietary Supplement: Placebo — single effect of placebo on muscular strength, power and endurance performance
  Arms: Placebo

SUMMARY:
Introduction: Several studies have evaluated and confirmed the ergogenic effect of acute caffeine and beetroot juice intake on sports performance. However, there are few studies focused on the production of strength, power, and muscle endurance, particularly when both supplements are ingested together.

Objectives: Evaluate the acute effect of combined and isolated intake of caffeine and beetroot juice on the production of strength, power, and muscle endurance in young adults, analyzing the effect of circadian rhythms (morning vs. afternoon) on the exercise performed (bench press vs. squat).

Methods: A total of 12 healthy and physically active participants will be recruited for the study. Through a double-blind, crossover, randomized, and controlled design, participants will ingest: a) Caffeine (3 mg/kg body mass); b) Beetroot juice (70 ml, 6.5 mmol of nitrates); c) Caffeine + Beetroot juice; d) Placebo (maltodextrin, 3 mg/kg). The supplements will be ingested 120 minutes (beetroot juice or placebo) and 60 minutes before (caffeine or placebo), the latter dissolved in 200 ml of water. After the ingestion period, strength, power, and muscle endurance will be analyzed with 1RM tests, strength and power tests at 25%, 50%, 75%, and 90% 1RM, and muscle endurance tests at 65% 1RM, in all cases for squat and bench press exercises. Additionally, dynamometry (manual and the isometric mid-thigh pull test) and vertical jump (squat jump and countermovement jump) will be analyzed. The four experimental conditions will be conducted in the morning (8:00 am to 10:00 am) and in the afternoon (4:30 pm to 6:30 pm).

ELIGIBILITY:
Inclusion Criteria:

* Age between ≥ 18 and ≤ 35 years.
* Body Mass Index (BMI) < 25 kg/m².
* Resistance-trained individuals (> 2 years of structured trained).
* Healthy men and women without neurological, cardiometabolic, immunological, or physical conditions that prevent them from exercising.
* Participants must be able to perform the tests described in the following section.

Exclusion Criteria:

* History of neuromuscular diseases, heart diseases, or diseases that may affect liver or muscle metabolism.
* Use of drugs, other stimulants or sport supplements that interfere with the intake of the study's dietary supplements.
* Sedentary habits (< 150 min/week of moderate exercise).
* Having undergone prolonged periods of forced physical inactivity during the 6 months prior to the study.
* Performing strenuous exercise during the 48 hours prior to the tests.
* Failure to replicate the same food intake on the two days of the experiments.
* Consuming caffeine or any other stimulant after 6 pm the day before the training or tests, to avoid headaches, discomfort, or lethargy among regular caffeine consumers.
* Consuming foods rich in NO3- (e.g., beetroot, spinach, or celery) during the 48 hours prior to each experimental condition.

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2024-01-30 (Actual); Study Completion 2024-05-01 (Actual)

PRIMARY OUTCOMES:
Mean and peak velocity and time to reach peak velocity at different %1RM | On each trial, after dietary supplement intake, during 2 weeks
  Measuring bar velocity desplacement during bench press and back squat exercises.
Mean and peak power output and time to reach peak power output at different %1RM | On each trial, after dietary supplement intake, during 2 weeks
  Measuring power output generated during bench press and back squat exercises.
Number of repetitions performed at 65%1RM until task failure | On each trial, after dietary supplement intake, during 2 weeks
  Additionally to mean and peak velocity, mean and peak power output, time to reach peak velocity and peak power

SECONDARY OUTCOMES:
Mood state (tension, depression, anger, vigor, fatigue and confusion) | On each trial, after dietary supplement intake, during 2 weeks
  Participants graded a set of 29 items related to the mood on a Likert scale from 0 (not at all) to 4 (extremely) in reply to the question "How do you feel at this moment?" to assess six scales: tension, depression, anger, vigor, fatigue and confusion.
Adverse effects | On each trial, after dietary supplement intake, during 2 weeks
  perception of power, endurance, energy and exertion, as well as heart, muscular and gastrointestinal discomfort.
handgrip and isometric mid-thigh pull tests | On each trial, after dietary supplement intake, during 2 weeks
  N generated
Vertical Jump (cm and power) | On each trial, after dietary supplement intake, during 2 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Facultad de Medicina y Ciencias de la Salud. Universidad de Alcalá, Alcalá de Henares, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Yes